CLINICAL TRIAL: NCT05736640
Title: The Effect of Denosumab on Periprosthetic Bone Mineral Density in Six Transfemoral Amputees Treated With Osseointegrated Implants: The Observations From a Terminated Randomized Controlled Trial
Brief Title: Osseointegrated Transdermal Femoral Amputation Prostheses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 34964
Record Dates: First submitted 2023-02-08; First posted 2023-02-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-02

CONDITIONS: Osseointegrated Implants; Bone Mineral Density
MeSH Terms: interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab (Active Comparator)
  Interventions: Drug: Denosumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Denosumab
  Arms: Denosumab
Drug: Placebo
  Arms: Placebo

SUMMARY:
Femur amputated patients often suffer from several problems with conventional socket prosthesis. Some experience changes in gait, discomfort when sitting, altered skin conditions (infection, irritation, rashes, sweat), phantom pain or lack of stabilization between the prosthesis and the residual limb. Many have a low score on "health-related quality of life" questionnaires (HRQL).

Some femur amputated patients may be a candidate to osseointegrated prosthesis. Osseointegrated prosthesis is an implant, where the fixture is inserted into the femur canal and an abutment screw, on which the leg-prostheses is inserted, protrudes the skin. By this procedure the patient have a high score on HRQL and experience fewer problems. They have improved gait, reduced discomfort when sitting, increased prosthetic use, and experience fewer skin and pain problems.

Femur amputee patients formerly mobilized on socket prosthesis have a reduced bone mineral density in the affected femur and pelvis.

The Phd-theses compromise of three studies. The aim of the first study is to follow patients with oosseointegrated prosthesis before and after surgery with DXA-scans to monitor the BMD. In the second study patients will be randomised to receive medical treatment with an RANKL-inhibitor, approved for treatment of osteoporosis, and monitored with DXA, microdialysis and radiostereometry. Depending on the DXA-results patients in the third study may receive fast track rehabilitation.

The hypothesis is that patients with osseointegrated prosthesis will have an increased BMD after surgery, 2 years follow up. Patients receiving RANKL inhibitor will have increased BMD, stability of the prosthesis, and some receive fast-track rehabilitation due to high BMD.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18-70 years
* Scheduled for OI-implant surgery
* Body mass index <30
* Female patients of childbearing age must produce a negative pregnancy test and use effective contraception
* informed consent

Exclusion Criteria:

* Diabetes with complication
* Atherosclerosis
* Smoking
* Drug abuse
* Treatment with NSAID or cytostatic
* Active cancer
* Liver or kidney insufficiency
* Dementia
* Hip flexion contracture on the affected side >10 degrees
* Body weight >100 kg
* Hypocalcaemia
* Contraindications to denosumab

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2016-09-20 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
change in periprosthetic bone mineral density | 30 months po